CLINICAL TRIAL: NCT07311083
Title: Feasibility of a Lifestyle Intervention to Switch to a High-fiber, Gut-healthy Diet in Women With Triple-negative Breast Cancer Undergoing Neoadjuvant Immunotherapy: a Randomized Controlled Trial
Brief Title: Feasibility of a Lifestyle Intervention for Women With Triple-negative Breast Cancer Under Neoadjuvant Immunotherapy
Acronym: BallastImmun
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kliniken Essen-Mitte (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024001-PV3
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Switching to a high-fibre diet in patients with TNBC undergoing neoadjuvant immunotherapy and chemot (Active Comparator): Switching to a high-fibre diet is supported by multi-professional consultation hours, individual counselling and group sessions that combine mind-body medicine and nutritional therapy content.
  Interventions: Other: switching to a high-fibre diet
- control group receives official dietary recommendations (Active Comparator): Control group receives standard care, i.e. a leaflet and an educational training video with dietary recommendations of the Deutsche Gesellschaft fuer Ernaehrung (DGE)
  Interventions: Other: official dietary recommendations

INTERVENTIONS:
Other: switching to a high-fibre diet — The aim of the intervention is to support patients in implementing a high-fibre diet (20-30 g of fibre per day) before and during systemic therapy. A multi-professional team consisting of a specialist doctor, a qualified nutritionist and an MBM therapist ensures comprehensive support during lifestyle modification. While the nutritional counselling provides recommendations for optimising diet, the MBM intervention addresses behavioural factors such as motivation, self-efficacy expectations and dealing with barriers to action. In addition, the specialist provides advice on symptom management.
  Arms: Switching to a high-fibre diet in patients with TNBC undergoing neoadjuvant immunotherapy and chemot
Other: official dietary recommendations — providing official dietary recommendations and an educational training video based on these recommendations of the guidelines of the German Nutrition Society (DGE)
  Arms: control group receives official dietary recommendations

SUMMARY:
Triple-negative breast cancer (TNBC) is considered a tumor with a high risk of recurrence and metastasis and requires aggressive systemic therapy combining immunotherapy and chemotherapy. If the therapy leads to complete remission (pCR), this is prognostically beneficial for patients.

Studies demonstrating the influence of the microbiome on the development of cancer and on the efficacy and toxicity of immunotherapy and chemotherapy underscore the potential of targeted nutritional interventions. Current data from microbiome research indicate that a high-fiber, gut-healthy diet modulates the microbiota in such a way that the response to and toxicity of immunotherapy and chemotherapy could be improved.

The aim of this project is to translate these findings into clinical care. The study will investigate whether an online integrative oncology group training program with mind-body elements supports and is feasible for the implementation of a high-fiber diet in patients with TNBC undergoing neoadjuvant immunotherapy and chemotherapy. The program will be compared with a control group that receives a flyer with nutritional recommendations. If the feasibility of this complementary medicine approach can be demonstrated, a confirmatory study is planned to investigate the expected effect on the pathological complete remission of TNBC.

DETAILED DESCRIPTION:
This study examines a nutritional concept developed specifically for this study with regard to the implementation of a switch to a high-fibre diet in patients with TNBC undergoing neoadjuvant immunotherapy and chemotherapy. This nutritional concept is embedded in an online, integrative oncology group training programme with mind-body medicine elements to support the change in diet and its tolerability. This intervention is compared with a control group that receives standard care, i.e. a flyer and an educational training video with nutritional recommendations based on the guidelines of the German Nutrition Society (DGE).

The following criteria have been established to determine the feasibility of these two target levels:

* Recruitment
* Consent to participate and randomisation
* Dropout rate
* Implementation of the intervention (dietary change and acceptance/effect of mind-body elements)
* Completeness of data collected for at least 80% of patients who complete the study

If the study proves feasible and demonstrates the viability of this integrative medical approach in women with TNBC undergoing neoadjuvant immunotherapy, a confirmatory intervention study with a larger sample size is planned. This study aims to contribute to expanding the current knowledge base and improving existing treatment options. The follow-up study aims to investigate the effects of the nutritional concept and the group training programme on the pCR of TNBC. It will analyse whether the nutritional concept and the group training programme enhance the response to immunotherapy and improve its tolerability in the study participants. The findings from this study will therefore be incorporated into the follow-up study, which will investigate the potential for an improved immune response to therapy and, at the same time, identify possible positive effects of the nutritional intervention on the side effect profile of immunotherapy. Furthermore, the design of the nutritional concept and/or the group training programme could be adapted for the follow-up study if the results are appropriate. The findings from both studies will then be transferred to clinical care, thereby optimising the current treatment options for TNBC patients and increasing their chances of recovery in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-75
* Histologically confirmed diagnosis of non-metastatic triple-negative breast cancer (TNM stage I-III) with planned neoadjuvant chemotherapy and immunotherapy
* Willingness to participate in the study and signed consent form

Exclusion Criteria:

* Advanced stage of disease with metastases
* Severe physical or psychopharmacologically treated psychiatric comorbidity that prevents a patient from participating in the study
* Pregnancy
* Participation in other clinical studies involving behavioral, psychological, or complementary medical interventions
* A diet that is incompatible with a high-fiber diet, such as the ketogenic diet
* Abuse of drugs and/or alcohol
* Inability to complete the questionnaires independently
* Colectomy
* Gastrointestinal stenosis
* Fructose intolerance
* Histamine intolerance
* Gluten intolerance
* Ketogenic diet
* Unwillingness to refrain from taking probiotics for the duration of the study
* Eating disorders
* No laptop and/or camera available to participate in the online group training program

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The primary target parameter is the feasibility of the planned study and the intervention. | from the enrolment to the end of treatment at 6.5 months
  The feasibility criteria are defined in the following categories: Recruitment:
  * Recruitment is considered feasible if the required sample size of n = 60 patients can be recruited within 17 months.
  * Randomisation: Randomisation is considered feasible if at least 25% of potentially eligible patients agree to participate in the study
  * Dropout rate: A maximum dropout rate of 20% per group is considered proof of feasibility.
  * Intervention: The intervention is considered feasible if at least 80% of the patients who complete the study are able to implement the nutritional intervention according to protocol. Implementation according to protocol is defined as a fibre intake of at least 20 g/day and the consumption of fermented foods.
  Data collection: Data collection is considered feasible if complete data on the planned primary endpoint parameter of the planned confirmatory study, pCR, is available for at least 80% of the patients who complete the study.

SECONDARY OUTCOMES:
Course of therapy (pCR) | 6 months after baseline
  Course of therapy in the sense of a complete response to systmatic therapy (= complete pathological remission)
Toxicity (CTCAE 6.0) including adverse events (AEs) | 6 months after baseline
  adverse events
Fatty acid profile (stool sample analysis) | baseline and 6 months after baseline
  Fatty acid profile
α-diversity and β-diversity of the microbiome (stool sample analysis) | baseline and 6 months after baseline
  diversity of the microbiome
Body weight | baseline, 1 to 3 weeks after baseline (start of the chemotherapy), 3 months after baseline, 6 months after baseline
  Body weight
Self-reported quality of life (FACT-B = Functional Assessment of Cancer Therapy - Breast) | baseline, 1 to 3 weeks after baseline (start of the chemotherapy), 3 months after baseline, 6 months after baseline
  quality of life, ranges from 0 to 4, with lower scores indicating higher stress levels which means a lower quality of life
Self-reported fatigue (FACIT fatigue = Functional Assessment of Chronic Illness Therapy Fatgigue) | baseline, 1 to 3 weeks after baseline (start of the chemotherapy), 3 months after baseline, 6 months after baseline
  Self-reported fatigue, scale from 0 to 4 with lower value indicating a greater fatigue. Two items are reversed.
Self-reported fiber intake (dietary records) | baseline, 1 to 3 weeks after baseline (start of the chemotherapy), 3 months after baseline, 6 months after baseline
  Self-reported fiber intake
Self-reported tolerance of increased fiber intake (IBS-SSS = irritable bowel syndrome severity scoring system) | baseline, 1 to 3 weeks after baseline (start of the chemotherapy), 3 months after baseline, 6 months after baseline
  Self-reported tolerance of increased fiber intake, symptoms are rated on a visual analog scale (VAS) from 0 to 100 points. 100 points indicate the most severe irritable bowel symptoms.
Adverse Events and Serious Adverse Events | baseline, 1 to 3 weeks after baseline (start of the chemotherapy), 3 months after baseline, 6 months after baseline
  Adverse Events and Serious Adverse Events